CLINICAL TRIAL: NCT07079449
Title: Trigger Point Injections for Myofascial Pain: A Comparative Study of Dry Needling, Lidocaine, and Mepivacaine
Brief Title: Comparison of Lidocaine, Mepivacaine, and Dry Needling in Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sümer Münevveroğlu (Other)
Responsible Party: Sponsor-Investigator, Sümer Münevveroğlu, Assistant Professor, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDIPOL-TMD-01
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Myofascial Pain Syndrome; Temporomandibular Joint Disorders; Facial Pain
Keywords: Trigger point injection; orofacial pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Temporomandibular Joint Disorders; Facial Pain | interventions — Dry Needling; Lidocaine; Mepivacaine

STUDY DESIGN:
Intervention Model Description: participants will be randomly assigned to one of three parallel arms: dry needling, lidocaine injection, or mepivacaine injection. All interventions will be applied once a week for three consecutive weeks. Outcome measures will be assessed at baseline and one week after the final injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine Group (Experimental): Participants in this group will receive lidocaine (20 mg/mL) injected into each bilateral active trigger point in the masseter and temporalis muscles once per week for three weeks.
  Interventions: Procedure: Lidocaine Hydrochloride
- Mepivacaine Group (Experimental): Participants in this group will receive mepivacaine (30 mg/mL) injected into each bilateral active trigger point in the masseter and temporalis muscles once per week for three weeks.
  Interventions: Procedure: Mepivacaine Hydrochloride
- Dry Needling Group (Experimental): Participants in this group will receive dry needling applied to bilateral active trigger points in the masseter and temporalis muscles. Treatment will be administered once a week for three weeks.
  Interventions: Procedure: Dry Needling

INTERVENTIONS:
Procedure: Dry Needling — Dry needling applied to bilateral active trigger points in the masseter and temporalis muscles once per week for three weeks.
  Arms: Dry Needling Group
Procedure: Lidocaine Hydrochloride — Lidocaine (20 mg/mL) injected into each active trigger point in the masseter and temporalis muscles once per week for three weeks.
  Arms: Lidocaine Group
Procedure: Mepivacaine Hydrochloride — Mepivacaine (30 mg/mL) injected into each active trigger point in the masseter and temporalis muscles once per week for three weeks.
  Arms: Mepivacaine Group

SUMMARY:
This randomized clinical trial will aim to compare the effectiveness of dry needling, lidocaine injection, and mepivacaine injection in the treatment of myofascial pain in the masticatory muscles. A total of 75 participants with bilateral active trigger points in the masseter and/or temporalis muscles will be enrolled and randomly assigned to three intervention groups. Each participant will receive weekly treatments for three weeks. Pain levels, depressive symptoms, and temporomandibular disorder severity will be assessed using the Visual Analog Scale, the Beck Depression Inventory, and the Fonseca Anamnestic Index. Outcome measures will be recorded at baseline and one week after the final treatment session. The primary objective of this study is to determine which intervention provides the greatest improvement in myofascial pain symptoms.

DETAILED DESCRIPTION:
This study will be a randomized, controlled clinical trial designed to compare the effectiveness of dry needling, lidocaine, and mepivacaine injections in the treatment of myofascial pain in the masticatory muscles. Seventy-five participants with bilateral active myofascial trigger points in the masseter and/or temporalis muscles will be recruited. Participants will be randomly assigned to one of three intervention groups: dry needling, lidocaine (20 mg/mL), or mepivacaine (30 mg/mL).

Injections will be administered once a week for three consecutive weeks to both sides of the face. Pain levels will be evaluated using the Visual Analog Scale, depressive symptoms with the Beck Depression Inventory and temporomandibular disorder severity with the Fonseca Anamnestic Index. Measurements will be performed at baseline (prior to first injection) and one week after the third and final injection.

The study will be conducted at Istanbul Medipol University with ethics committee approval. Participants will be informed about the study procedures and informed consent will be obtained from all subjects. The primary objective of the study is to evaluate which intervention provides the most significant reduction in pain and associated symptoms of myofascial pain syndrome. Secondary outcomes will include improvements in depressive symptoms and temporomandibular disorder-related limitations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 64 years
* Presence of bilateral active myofascial trigger points in both the masseter and temporalis muscles
* Pain provoked by approximately 1 kg of external digital pressure on trigger points
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Previous or ongoing treatment for temporomandibular disorders (e.g., occlusal splints, botulinum toxin injections)
* Presence of systemic neuromuscular disease
* Pregnancy or breastfeeding
* Use of analgesics, muscle relaxants, or antidepressants within the past 2 weeks
* Active infection, tumor, or trauma in the orofacial region

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity based on the Visual Analog Scale | Baseline and one week after the third injection
  Pain intensity will be assessed using a 10 cm Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates the worst possible pain. The change in VAS scores from baseline to post-treatment will be analyzed.

SECONDARY OUTCOMES:
Change in depressive symptoms based on the Beck Depression Inventory | Baseline and one week after the third injection
  Change in depressive symptoms based on the Beck Depression Inventory (BDI). The BDI is a 21-item self-reported questionnaire that measures depressive symptoms. Scores range from 0 to 63, with higher scores indicating more severe depression.
Change in temporomandibular disorder severity based on the Fonseca Anamnestic Index | Baseline and one week after the third injection
  Change in temporomandibular disorder severity based on the Fonseca Anamnestic Index.
  The Fonseca Anamnestic Index consists of 10 items assessing TMD-related symptoms. Total scores range from 0 to 100, with higher scores indicating more severe temporomandibular dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No